CLINICAL TRIAL: NCT03096717
Title: Incidence of Dysplasia and Colorectal Cancer in Patients With Chronic Idiopathic Inflammatory Colitis Treated With Biologics, Mesalamine, and Immunosuppressive Drug Combinations
Brief Title: Dysplasia in Inflammatory Chronic Idiopathic Colitis Long-standing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, alba panarese, principal investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 7
Record Dates: First submitted 2017-03-26; First posted 2017-03-30 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Dysplasia in IBD
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — colonic biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: colonoscopy and histology — colonic biopsies for detection of dysplasia

SUMMARY:
Chronic intestinal inflammation produce dysplasia more frequently than the normal population. The therapies protect against these changes, but do not rule out dysplasia. It is not known the effect of different therapies protection.

DETAILED DESCRIPTION:
The literature data show that the inflammatory bowel diseases (rectal ulcerative colitis and Crohn's disease) determine an increased risk of developing dysplasia and cancer of the colon and rectum, for the chronic inflammation that they fee, with the differences that the two diseases arise. The progression from normal mucosa to dysplasia and then to cancer is more rapid than in the adenoma-carcinoma sequence.

In patients with idiopathic chronic inflammatory colitis drug therapies in use reduce the incidence of dysplasia.

A systematic review concluded in favor of a chemo preventive effect of mesalazine. In any case, it has been reported protective association between use of mesalazine and cancer associated with colitis (colitis Associated carcinoma CAC) with an odds ratio of 0.51 per CAC / dysplasia. This data, in subsequent studies, including recent ones, have remained controversial.

The introduction of biological drugs in the treatment of patients with inflammatory bowel disease (IBD) has changed the quality of life and also the natural history of the disease. It is not known what biological drugs have improved the clinical history of these diseases by changing the incidence of dysplasia and colorectal cancer.

The treatment of idiopathic inflammatory bowel diseases (IBD), the last decade has seen profound changes and, now, the use of biological drugs is frequent in the moderate-severe forms, especially if extended. Mesalazine has in the indication of mild to moderate forms of therapy.

ELIGIBILITY:
Inclusion Criteria:

* long standing colonic inflammatory bowel disease
* clinical, endoscopic and histological remission
* completeness of data

Exclusion Criteria:

* important comorbidities
* family history of colorectal cancer
* insufficient data

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with long standing idiopathic chronic colitis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-01-21 (Estimated)

PRIMARY OUTCOMES:
incidence of dysplasia in relation to therapy performed | 24 months
  colonic biopsies are performed in long standing inflammatory bowel disease in relation to dysplasia detection in patients on different drugs therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Alba Panarese, Castellana Grotte, Apulia, Italy

IPD SHARING:
Plan to Share IPD: Yes